CLINICAL TRIAL: NCT04599764
Title: High Definition Transcranial Direct Current Stimulation (HD-tDCS) for Early Alzheimer's Disease
Acronym: HD-tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AH med university2018913
Record Dates: First submitted 2020-10-18; First posted 2020-10-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Transcranial Direct Current Stimulation; Functional Magnetic Resonance Imaging; Early Alzheimer's Disease
Keywords: High Definition Transcranial Direct Current Stimulation; Functional Magnetic Resonance Imaging; Neuropsychology; Early Alzheimer's Disease; Working Memory; Alzheimer's Disease Assessment Scale-Cognitive Subscale
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Caregivers, subjects, and evaluators remain blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham-Anode tDCS&Cognitive training (Sham Comparator): Participants will receive Cognitive training+Sham tDCS daily for two weeks
  Interventions: Other: computer-based cognitive training; Other: Sham tDCS
- Anodal tDCS with Cognitive training (Active Comparator): Participants will receive anoale tDCS daily and cognitive training for two weeks
  Interventions: Other: HD-tDCS; Other: computer-based cognitive training
- Anodal tDCS without Cognitive training (Active Comparator): Participants will receive anoale tDCS daily without cognitive training for two weeks
  Interventions: Other: HD-tDCS

INTERVENTIONS:
Other: HD-tDCS — Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation tool that alters cortical excitability and activity via application of weak direct currents.HD-tDCS was administered using the Soterix 1×1 tDCS Low-Intensity Stimulator and the Soterix 4×1 Adapter. The selection of the electrode montage was based on computational models generating simulated current topography using HD Explore, which demonstrated good current distribution in the left dorsolateral prefrontal cortex (DLPFC). For left DLPFC stimulation, the anodal electrode was placed at the F3 position (using the International 10-20 EEG system), and the 4 return electrodes (cathodes) were placed at positions AFz, FCz, F7, and C5 (4-6 cm from the anode). The center position CZ was aligned with the vertex of the head. During anodal DLPFC stimulation, participants received stimulation at 2 mA for 30 minutes, including a 30-second ramp-up period at the start and a 30-second ramp-down period at the end.
  Arms: Anodal tDCS with Cognitive training; Anodal tDCS without Cognitive training
Other: computer-based cognitive training — Computer-based cognitive training (CCT) is a potentially important tool for individuals at risk of dementia. This trial will employ a computerized multi-domain adaptive training program. This program and training model have been demonstrated to be effective and beneficial in patients with vascular cognitive impairment. In the CCT intervention group, participants will undergo 2 weeks of computerized, multi-domain, adaptive training. The training domains include processing speed, attention, perception, long-term memory, working memory, calculation, executive control, reasoning, and problem-solving. Task rigor varies across domains and determines task grouping. Participants are required to complete 30 minutes of daily training(one session each of six 5-minute tasks).
  Arms: Anodal tDCS with Cognitive training; Sham-Anode tDCS&Cognitive training
Other: Sham tDCS — Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation tool that alters cortical excitability and activity via application of weak direct currents.HD-tDCS was administered using the Soterix 1×1 tDCS Low-Intensity Stimulator and the Soterix 4×1 Adapter. The selection of the electrode montage was based on computational models generating simulated current topography using HD Explore, which demonstrated good current distribution in the left dorsolateral prefrontal cortex (DLPFC). For left DLPFC stimulation, the anodal electrode was placed at the F3 position (using the International 10-20 EEG system), and the 4 return electrodes (cathodes) were placed at positions AFz, FCz, F7, and C5 (4-6 cm from the anode). The center position CZ was aligned with the vertex of the head. For sham stimulation, participants received only the initial 30-second ramp-up to 2 mA, after which stimulation was immediately terminated.
  Arms: Sham-Anode tDCS&Cognitive training

SUMMARY:
To investigate the clinical effect neural mechanism of high-definition transcranial direct current stimulation combined with cognitive training on early AD

DETAILED DESCRIPTION:
Upon meeting the inclusion criteria and providing informed consent, each participant will complete a series of cognitive assessments and tDCS at the hospital outpatient clinics or inpatient department. Participants were randomly allocated to anode tDCS group with cognitive training, anode tDCS group and the sham group. There are about 20 participants in each group. Participants were studied using a double-blind design. Study participants and all personnel responsible for the effects of the participants remained masked to allocated condition and allocation parameters. Only tDCS administrators had access to the randomization list; they had minimal contact with the participants, and no role in cognitive assessments. For the first 30 participants, allocation was decided by draw. For the subsequent 30 patients, allocation was according to computer generated random numbers. Each participant would be treated for 10 days in two weeks by HD-tDCS.

Before the tDCS, a series of cognitive assessments and neuropsychological tests were obtained by a trained investigator to assess baseline. Each assessment will involve a set of assessment tools, including Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog), Montreal Cognitive Assessment (MoCA) and associative memory as the primary outcome measure and various other tasks and questionnaires to measure cognition(DS, Stroop test, VFT, SDMT), memory (AVLT, AMT, working memory test), emotion(HAMA-17, HAMD-14, eye-tracking technolodgy), executive function(SST, WSCT, GDT) and stimulation tolerability. All the tests are conducted in two days. The participants had receiving a magnetic resonance imaging scan in multi-modalities, and electroencephalography (EEG) record.

Evaluations were conducted one week after treatment and at the end of two weeks of treatment, as well as the Global Index of Safety to assess adverse events of the stimulation. Participants were instructed to focus their answers on the past 7/14 days. The participants had also receiving a battery measure of neuropsychological tests, magnetic resonance imaging scan in multi-modalities, and EEG record. All tests were instructed to finished within 24 hours after the last stimulation. One month and three months after the last stimulation, participants were interviewed to obtain the same assessment as before. They were instructed to focus their answers on the past months.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with early Alzheimer's disease or related diseases according to NINCDS-ACDRADA criteria.
* Subjects must have a MMSE score between 10 and 27,indicating mild cognitive impairment or dementia
* CDR score ≤ 2
* Subject under treatment by IAChE for at least 3 months.
* psychotropic treatments are tolerated if they were administered and unchanged for at least 3 months

Exclusion Criteria:

* CDR > 2
* Any history or clinical signs of other severe psychiatric illnesses (like major depression,psychosis or obsessive compulsive disorder).
* History of head injury,stroke,or other neurologic disease.
* Organic brain defects on T1 or T2 images.
* History of seizures or unexplained loss of consciousness.
* Implanted pacemaker,medication pump,vagal stimulator,deep brain stimulator.
* Family history of medication refractory epilepsy.
* History of substance abuse within the last 6 months.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Memory improved assessed by Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | changes from baseline at 7,14 days and 4,12 weeks post-treatment
  This is an very common clinical motor estimating scale. including orientation, language, structure, application of concepts, immediate recall of words and recognition of words, with a full score of 70. Higher scores indicate worse symptoms.

SECONDARY OUTCOMES:
special-version working memory | changes from baseline at 7,14 days and 4,12 weeks post-treatment
  the accuracy and reaction time in working memory task
Associative Memory | changes from baseline at 7,14 days and 4,12 weeks post-treatment
  The changes in Associative Memory will constitute the major research outcome measure used to assess response to HD-tDCS.
MMSE(Mini Mental State Examination) | changes from baseline at 7,14 days and 4,12 weeks post-treatment
  The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better.
LMT (Logic Memory Test) | changes from baseline at 7,14 days and 4,12 weeks post-treatment
  The changes in LMT will constitute the secondary research outcome

OTHER OUTCOMES:
DST (Digital Span Test; Forward and Backward) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The changes in DST will constitute the other research outcome.
TMT (Trail Making Test) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The Trail Making Test (TMT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.
HAMD (Hamilton Depression Scale) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The changes in HAMD will constitute the other research outcome. The examination content consists of 17 questions (about 10 minutes), with a full score of 52. The higher the score, the more severe the depressive symptoms are.
HAMA (Hamilton Anxiety Scale) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The changes in HAMD will constitute the other research outcome. The examination content consists of 14 questions (about 10 minutes), with a full score of 56. The higher the score, the more severe the anxiety symptoms are.
NPI (Neuropsychiatric Inventory) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The changes in HAMD will constitute the other research outcome.
MRI measures | changes from baseline at 14 days and 4,12 weeks post-treatment
  Multimodal magnetic resonance data were acquired, including structural phase magnetic resonance and rest state magnetic resonance.
changes in Montreal Cognitive Assessment (MoCA) | changes from baseline at 14 days and 4,12 weeks post-treatment
  MoCA was developed by Nasreddine et al. based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. We adopted a localized version (Mandarin version，includes 2 alternative versions) in line with the Chinese cultural background.It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score.
GDS(Geriatric depression scale) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The Geriatric Depression Scale (GDS) was created in 1982 by Brank et al. and is dedicated to screening for depression in the elderly. The most suitable feelings for the elderly in the past week were evaluated.There are 30 items in the scale, the total score is 30 points. The higher the score, the more obvious the depressive symptoms. It is generally considered that less than 10 points is normal.
JLOT(Judgment of line Judgment of line orientation test orientation test) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The JLOT test was determined by Benton et al. in 1994. There are two versions of H and V. The difference is that the order in which the pictures are presented is different. Each version contains 35 images, of which the official test consists of 30 images, and the other 5 images are for the participants to learn. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.
HVOT(Hooper visual organization test Hooper visual organization test) | changes from baseline at 14 days and 4,12 weeks post-treatment
  The changes in HVOT(Hooper visual organization test Hooper visual organization test) will constitute assess response to rTMS the secondary research outcome measure.HVOT is a cognitive test used to evaluate the perceived structure of the subject. It consists of 30 items，and each question is 1 point and the total score is 30 points. The final score is the correct number of subjects to answer, the full score is 30 points, the higher the score, the better the space perception ability of the subject.
The Stroop color test | changes from baseline at 14 days and 4,12 weeks post-treatment
  The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China